CLINICAL TRIAL: NCT00700401
Title: A Prospective, Observational Study to Assess the Virological Response at Week 4 to the Therapy With PEGASYS® (Peginterferon Alfa 2a) Plus COPEGUS® (Ribavirin) in a Population of Treatment Naïve Patients With Chronic Hepatitis C, Genotype 2 or 3.
Brief Title: POTENTE Study: A Study of Early Virological Response in Naive Patients With Chronic Hepatitis C, Genotype 2 or 3, Treated With PEGASYS (Peginterferon Alfa-2a (40KD)) Plus Copegus (Ribavirin).
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21543
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Results first posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-05

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Peginterferon Alfa-2a + Ribavirin
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin [Copegus]

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — 180 micrograms/week sc for 24 weeks
Drug: ribavirin [Copegus] — 800mg po daily for 24 weeks

SUMMARY:
This single arm study will investigate the predictive value of a week 4 virological response on sustained virological response in patients with chronic hepatitis C, genotype 2 or 3, treated with PEGASYS + Copegus. Eligible patients will be treated with PEGASYS 180 micrograms/week sc + Copegus 800mg/day po; those who have a virological response at week 4 will continue to be treated for 24 weeks, followed by a 24 week treatment-free follow-up. Non-responders at week 4 will be entered into a separate protocol (MV21371) to receive PEGASYS + Copegus for 24 or 48 weeks. The anticipated time on study treatment is 3-12 months, and the target sample size is 100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* positive serum HCV RNA.

Exclusion Criteria:

* co-infection with HIV or HBV (patients with a positive HBsAg);
* previous treatment with interferon, or peginterferon and/or ribavirin;
* severe hepatic dysfunction or decompensated cirrhosis of liver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with serologically proven chronic hepatitis C and genotype 2 or 3, with or without cirrhosis and compensated liver disease (Child-Pugh A cirrhosis.)
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2008-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Brazil (10):
  - Vitória, Espírito Santo
  - Brasília, Federal District
  - São Luís, Maranhão
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - Campinas, São Paulo
  - Ribeirão Preto, São Paulo
  - Santo André, São Paulo
  - São Paulo, São Paulo
  - Sorocaba, São Paulo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 262 participants were enrolled from 13 centers in Brazil. This study was conducted between 26 November 2008 and 19 November 2010.
Groups:
- Peginterferon Alfa-2a + Ribavirin: Eligible participants receiving peginterferon alfa-2a (Pegasys) 180 microgram (µg) subcutaneously once a weekly with ribavirin (Copegus) 800 mg or 1000/1200 mg/day, according to the body weight (1000 mg [<75kg] or 1200 mg [>/=75 kg]) for 24 weeks were observed.
Period: Overall Study
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Started | 262
Completed | 168
Not Completed | 94
Not completed — Detectable HCV RNA after Week 4 | 82
Not completed — Adverse Event | 5
Not completed — Refused Treatment | 2
Not completed — Lost to Follow-up | 1
Not completed — Treatment never started | 1
Not completed — HCV RNA not detected at baseline and SAE | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population included all participants who received at least one dose of study drug.
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 262
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118
  Male | 144

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virological Response at Week 48
Description: Sustained Virological Response (SVR) is defined as participants with undetectable Hepatitis C Virus (HCV) ribonucleic acid (RNA) at 24 weeks after the last dose of study drug. The detection limit of HCV RNA was 15 international units (IU) per milliliter (mL) by qualitative polymerase chain reaction (PCR).
Time Frame: At Week 48
Population: Intention-to-treat (ITT) population included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 262
Percentage of participants | 52.7 [46.6 to 58.6]

2. Secondary Outcome: Percentage of Participants With Rapid Virological Response at Week 4
Description: Rapid Virological Response (RVR) is defined as participants with) undetectable HCV RNA at 4 weeks after initiation of the treatment period. The detection limit of HCV RNA was 15 IU/mL by qualitative PCR.
Time Frame: At Week 4
Population: Intention-to-treat (ITT) population included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 262
Percentage of participants | 56.9 [50.8 to 62.7]

3. Secondary Outcome: Percentage of Participants With Virological Response at Week 24
Description: Virological response is defined as participants with undetectable HCV RNA after the last dose of study drug (Week 24).
Time Frame: At Week 24
Population: Intention-to-treat (ITT) population included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 262
Percentage of participants | 56.9 [50.8 to 62.7]

4. Secondary Outcome: Percentage of Participants With Virological Relapse
Description: Virological relapse is defined as participants with virological response (undetectable HCV RNA) but did not achieve SVR.
Time Frame: At week 48
Population: Intention-to-treat (ITT) population included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 149
Percentage of participants | 9.4 [5.7 to 15.2]

5. Secondary Outcome: Percentage of Participants With Positive Predictive Value
Description: Positive predictive value is defined as participants with RVR who did not achieve SVR.
Time Frame: At Week 48
Population: Intention-to-treat (ITT) population included all participants who received at least one dose of study drug. Data of participants available at the assessment time point were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 149
percentage of participants | 85.2 [78.7 to 90.0]

6. Secondary Outcome: Number of Participants With Any Adverse Events and Any Serious Adverse Events
Description: An any adverse events (AEs) is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. An serious adverse events (SAEs) is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect.
Time Frame: Up to 48 weeks
Population: Intention-to-treat (ITT) population included all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 262
participants
  Any AEs | 196
  Any SAEs | 13

7. Secondary Outcome: Mean Percent Change From Baseline in Hematology Parameters at Weeks 2, 4, 12, 24, and 48
Description: Hematology parameters included hemoglobin, hematocrit, leukocytes, neutrophils and platelets.
Time Frame: At Baseline (Day 0), Week 2, Week 4, Week 12, Week 24 and Week 48
Population: Intention-to-treat (ITT) population included all participants who received at least one dose of study drug. Data of participants available at the assessment time point were included in the analysis. 'n' is number of participants analyzed at the specified weeks.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 259
Percent change
  Hemoglobin, Week 2 ( n =257) | -8.4 (0.5)
  Hemoglobin, Week 4 (n=259) | -15.7 (0.6)
  Hemoglobin, Week 12 (n=157) | -19.6 (0.7)
  Hemoglobin, Week 24 (n=156) | -20.7 (0.8)
  Hemoglobin, Week 48 (n=110) | -2.2 (0.6)
  Hematocrit, Week 2 ( n = 255) | -8.1 (0.5)
  Hematocrit, Week 4 (n = 257) | -14.5 (0.5)
  Hematocrit, Week 12 (n = 156) | -17.7 (0.7)
  Hematocrit, Week 24 (n = 155) | -17.9 (0.8)
  Hematocrit, Week 48 (n=110) | -2.3 (0.6)
  Leukocytes, Week 2 ( n = 256) | -33.2 (1.2)
  Leukocytes, Week 4 (n = 258) | -43.4 (1)
  Leukocytes, Week 12 (n = 157) | -48.1 (2.1)
  Leukocytes, Week 24 (n = 156) | -52.1 (1.4)
  Leukocytes, Week 48 (n = 110) | 0.3 (2.5)
  Neutrophils, Week 2 ( n = 256) | -42.9 (2.4)
  Neutrophils, Week 4 (n = 258) | -48 (2.5)
  Neutrophils, Week 12 (n = 157) | -47.3 (4.1)
  Neutrophils, Week 24 (n = 156) | -53.6 (2)
  Neutrophils, Week 48 (n = 110) | 4.5 (3.7)
  Platelets, Week 2 ( n = 257) | -18.3 (1.7)
  Platelets, Week 4 (n = 259) | -20.4 (1.5)
  Platelets, Week 12 (n = 157) | -26.7 (2.4)
  Platelets, Week 24 (n = 155) | -27.6 (1.9)
  Platelets, Week 48 (n = 110) | 4 (4.3)

8. Secondary Outcome: Mean Percent Change From Baseline in Biochemistry Parameters at Weeks 4, 12, 24 and 48
Description: Biochemistry parameters included alanine transaminase (ALT), aspartate transaminase (AST), gamma-glutamyl transpeptidase (Gamma-GT),fasting cholesterol, blood glucose, insulin, total bilirubin, creatinine, triglycerides, homeostatic model assessment score, prothrombin time (PT) and international normalized ratio (INR). The homeostatic model assessment (HOMA) score is a method used to quantify insulin resistance. HOMA score = (fasting glucose in mg/dL × fasting insulin in μIU/mL) / 405. A normal participant can have a HOMA score up to 3. A patient with a score of >3 is definitely insulin resistance. Low HOMA score indicate high insulin resistance, whereas high HOMA score indicate low insulin resistance.
Time Frame: Baseline, Week 4, Week 12, Week 24 and Week 48
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 257
Percent change
  ALT, Week 4 ( n = 257) | -28.5 (4.8)
  ALT, Week 12 (n = 159) | -30.4 (5.5)
  ALT, Week 24 (n = 156) | -30 (8.6)
  ALT, Week 48 (n = 125) | -61.8 (3.1)
  AST, Week 4 ( n = 256) | -19.6 (2.7)
  AST, Week 12 (n = 159) | -10.2 (4.9)
  AST, Week 24 (n = 156) | -7.6 (8.4)
  AST, Week 48 (n = 125) | -47.2 (2.9)
  Gamma-GT, Week 4 ( n = 243) | 11.8 (3.3)
  Gamma-GT, Week 12 (n = 151) | 32.5 (7.9)
  Gamma-GT, Week 24 (n = 149) | 69.2 (25.3)
  Gamma-GT, Week 48 (n = 121) | -33.4 (3.5)
  Fasting cholesterol, Week 4 ( n = 214) | -1 (1.6)
  Fasting cholesterol, Week 12 (n = 130) | -1.4 (2.4)
  Fasting cholesterol, Week 24 (n = 123) | 0.6 (2.7)
  Fasting cholesterol, Week 48 (n = 97) | 15.6 (2.7)
  Fasting blood glucose, Week 4 ( n = 229) | -3.5 (1.1)
  Fasting blood glucose, Week 12 (n = 135) | -1.8 (2.5)
  Fasting blood glucose, Week 24 (n = 136) | 1.3 (2.4)
  Fasting blood glucose, Week 48 (n = 111) | -1.2 (2.1)
  Fasting insulin, Week 4 ( n = 131) | 22.9 (11.3)
  Fasting insulin, Week 12 (n = 79) | 11.1 (11.6)
  Fasting insulin, Week 24 (n = 74) | -12.2 (5.8)
  Fasting insulin, Week 48 (n = 68) | 18.3 (16.7)
  Total bilirubin, Week 4 ( n = 234) | 32.8 (4.4)
  Total bilirubin, Week 12 (n = 148) | 19.3 (5.3)
  Total bilirubin, Week 24 (n = 123) | 0 (3.9)
  Total bilirubin, Week 48 (n = 108) | -1.7 (4.5)
  Creatinine, Week 4 ( n = 239) | -1.82 (0.99)
  Creatinine, Week 12 (n = 138) | -2.71 (1.43)
  Creatinine, Week 24 (n = 133) | -3.55 (1.55)
  Creatinine, Week 48 (n = 116) | 5.89 (1.78)
  Fasting triglycerides, Week 4 ( n = 212) | 44.7 (4.8)
  Fasting triglycerides, Week 12 (n = 128) | 56 (7.2)
  Fasting triglycerides, Week 24 (n = 121) | 58.1 (7.3)
  Fasting triglycerides, Week 48 (n = 92) | 22 (6.5)
  HOMA score, Week 4 ( n = 46) | 12.6 (23.3)
  HOMA score, Week 12 (n = 37) | 10.3 (20.6)
  HOMA score, Week 24 (n = 28) | -14.6 (11.6)
  HOMA score, Week 48 (n = 20) | 10.9 (19.3)
  PT, Week 4 ( n = 55) | -1.9 (0.7)
  PT, Week 12 (n = 31) | -2.6 (1)
  PT, Week 24 (n = 26) | -3.5 (1.7)
  PT, Week 48 (n = 30) | -4.1 (1)
  INR, Week 4 ( n = 151) | 0.1 (1.3)
  INR, Week 12 (n = 73) | -1.1 (0.8)
  INR, Week 24 (n = 73) | -1.5 (1.1)
  INR, Week 48 (n = 71) | -3.2 (0.8)

ADVERSE EVENTS:
Time Frame: Up to 48 weeks
Description: Serious adverse events (SAEs) and non-serious AEs were reported for the safety population which included all participants who received at least one dose of study drug.
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Serious Adverse Events (participants affected / at risk) | 13/262
Other Adverse Events (participants affected / at risk) | 179/262
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a + Ribavirin (N=262)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 1
Anorectal operation (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Cellulitis (Infections and infestations) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Pneumonia (Infections and infestations) | 1
Salivary gland mass (Gastrointestinal disorders) | 1
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a + Ribavirin (N=262)
Anaemia (Blood and lymphatic system disorders) | 27
Neutropenia (Blood and lymphatic system disorders) | 18
Nausea (Gastrointestinal disorders) | 27
Pyrexia (General disorders) | 51
Asthenia (General disorders) | 42
Fatigue (General disorders) | 32
Influenza like illness (General disorders) | 23
Irritability (General disorders) | 20
Pain (General disorders) | 16
Decreased appetite (Metabolism and nutrition disorders) | 42
Myalgia (Musculoskeletal and connective tissue disorders) | 42
Arthralgia (Musculoskeletal and connective tissue disorders) | 17
Headache (Nervous system disorders) | 69
Insomnia (Nervous system disorders) | 19
Depression (Psychiatric disorders) | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Pruritus (Skin and subcutaneous tissue disorders) | 30
Alopecia (Skin and subcutaneous tissue disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.